CLINICAL TRIAL: NCT00949533
Title: A Phase IIIb, Open-label, Comparative, Randomized Study on Resistance of Influenza A/H1N1 2009 Virus to Treatment With Oseltamivir at Standard Dose Versus Double Dose
Brief Title: A Study on Emergence of Resistance With Oseltamivir (Tamiflu) in Participants With Seasonal Influenza
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML22789
Record Dates: First submitted 2009-07-15; First posted 2009-07-30 (Estimated); Results first posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-06

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

ARMS (2):
- Standard Dose (Experimental): Oseltamivir capsule will be administered orally at a dose of 75 mg BID in adult participants and children will receive oseltamivir powder for oral suspension dose (at 12 milligrams/ milliliter [mg/mL]) based on their body weight with a starting dose of 30 mg BID to a maximum dose of 75 mg BID; for 5 days.
  Interventions: Drug: Oseltamivir
- Double Dose (Active Comparator): Oseltamivir capsule will be administered orally at a dose of 150 mg BID in adult participants and children will receive oseltamivir powder for oral suspension dose (at 12 mg/mL) based on their body weight with a starting dose of 60 mg BID to a maximum dose of 150 mg BID; for 5 days.
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Oseltamivir — Standard dose (30 - 75 mg orally bid) or double dose (60 - 150 mg orally bid); for 5 days
  Other Names: Tamiflu

SUMMARY:
This open-label randomized 2 arm study will determine the emergence of viral resistance in participants with seasonal influenza A infection treated with oseltamivir. Eligible participants less than or equal to (</=) 5 years of age will be randomized to receive oseltamivir at either standard dose (30-75 milligrams [mg] orally twice daily [bid]) or double dose (60-150 mg orally bid) for 5 days. Target sample size is greater than (>) 100.

ELIGIBILITY:
Inclusion Criteria:

* positive rapid antigen test for influenza A
* onset of symptoms of influenza (fever, at least one respiratory symptom) </=48 hours

Exclusion Criteria:

* clinical suspicion of infection with a respiratory virus other than influenza
* suspicion of invasive bacterial infection
* evidence of poorly controlled underlying disease
* known immunosuppression
* known allergy to Oseltamivir
* women who are pregnant or planning to get pregnant during the study

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Brazil (2):
  - Curitiba
  - São Paulo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 199 participants, 162 were considered as screening failures, mainly due to the negative result detected by the quick test for Influenza A Antigen. Therefore, 37 participants included in the study.
Groups:
- Standard Dose: Oseltamivir (Tamiflu) capsule was administered orally at a dose of 75 milligrams (mg) twice a day (BID) in adult participants and children received oseltamivir powder for oral suspension dose (at 12 milligrams/ milliliter [mg/mL]) based on their body weight with a starting dose of 30 mg BID to a maximum dose of 75 mg BID; for 5 days.
- Double Dose: Oseltamivir capsule was administered orally at a dose of 150 mg BID in adult participants and children received oseltamivir powder for oral suspension dose (at 12 mg/mL) based on their body weight with a starting dose of 60 mg BID to a maximum dose of 150 mg BID; for 5 days.
Period: Overall Study
Arm/Group | Standard Dose | Double Dose
Started | 19 | 18
Completed | 19 | 17
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population included all enrolled participants who received at least one dose of the study drug.
Groups:
- Standard Dose: Oseltamivir capsule was administered orally at a dose of 75 mg BID in adult participants and children received oseltamivir powder for oral suspension dose (at 12 mg/mL) based on their body weight with a starting dose of 30 mg BID to a maximum dose of 75 mg BID; for 5 days.
- Total: Total of all reporting groups
Arm/Group | Standard Dose | Double Dose | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.6 (11.0) | 22.0 (12.7) | 21.8 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Excreting Resistant Virus
Description: Resistant virus included new influenza A virus subtype hemagglutinin type 1 and neuraminidase type 1 (New AH1N1).
Time Frame: Day 5
Population: ITT population. Here "number of participants analyzed" included evaluable participants for the outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Standard Dose | Double Dose
Number analyzed (Participants) | 19 | 17
percentage of participants | 26.3 | 35.3
Statistical Analysis 1: Comparison: Standard Dose vs Double Dose; Test type: Superiority or Other; p = 0.825, Pearson Chi-Square

2. Secondary Outcome: Percentage of Participants With A Reduction in Viral Load
Description: Viral load is defined as the amount of H1N1 virus in blood. As per investigator, a participant was considered as having viral load reduction at Day 5 if the Day 5 viral load was lower than the Baseline viral load.
Time Frame: Baseline, Day 5
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Standard Dose | Double Dose
Number analyzed (Participants) | 19 | 18
percentage of participants | 100 | 100
Statistical Analysis 1: Comparison: Standard Dose vs Double Dose; Test type: Superiority or Other; p > 0.05, Chi-squared

3. Secondary Outcome: Number of Participants With Various Clinical Signs and Symptoms
Description: Number of participants with various clinical signs and symptoms, as per investigator's discretion, were reported. Same participants were reported in more than 1 category. "Other" in the category included abdominal pain, breathlessness, thoracic pain and tired.
Time Frame: Day 5
Population: ITT population. Here "number of participants analyzed" included evaluable participants for the outcome measure.
Measure: Number; unit: participants
Arm/Group | Standard Dose | Double Dose
Number analyzed (Participants) | 19 | 17
participants
  Cough | 10 | 9
  Rhinorrhea | 10 | 5
  Sore throat | 2 | 2
  Shortness of breath | 2 | 1
  Diarrhea | 2 | 0
  Headache | 1 | 2
  Conjunctivitis | 1 | 0
  Vomiting | 1 | 0
  Other | 4 | 0
Statistical Analysis 1: Comparison: Standard Dose vs Double Dose; Cough: statistical difference between 2 groups was based on chi-squared test; Test type: Superiority or Other; p = 1.000, Chi-squared
Statistical Analysis 2: Comparison: Standard Dose vs Double Dose; Rhinorrhea: statistical difference between 2 groups was based on chi-squared test; Test type: Superiority or Other; p = 0.284, Chi-squared
Statistical Analysis 3: Comparison: Standard Dose vs Double Dose; Sore throat: statistical difference between 2 groups was based on fisher-exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 4: Comparison: Standard Dose vs Double Dose; Shortness of breath: statistical difference between 2 groups was based on fisher-exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 5: Comparison: Standard Dose vs Double Dose; Diarrhea: statistical difference between 2 groups was based on fisher-exact test; Test type: Superiority or Other; p = 0.487, Fisher Exact
Statistical Analysis 6: Comparison: Standard Dose vs Double Dose; Headache: statistical difference between 2 groups was based on fisher-exact test; Test type: Superiority or Other; p = 0.593, Fisher Exact
Statistical Analysis 7: Comparison: Standard Dose vs Double Dose; Conjunctivitis: statistical difference between 2 groups was based on fisher-exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 8: Comparison: Standard Dose vs Double Dose; Vomiting: statistical difference between 2 groups was based on fisher-exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 9: Comparison: Standard Dose vs Double Dose; Other: statistical difference between 2 groups was based on fisher-exact test; Test type: Superiority or Other; p = 0.106, Fisher Exact

4. Secondary Outcome: Number of Participants With Various Clinical Signs and Symptoms in Whom Resistant Virus Were Detected
Description: Number of participants with various clinical signs and symptoms, as per investigator's discretion, in whom new AH1N1 virus was detected, were reported. Same participants were reported in more than 1 category.
Time Frame: Day 5
Population: ITT population. Here "number of participants analyzed" included evaluable participants for the outcome measure.
Measure: Number; unit: participants
Arm/Group | Standard Dose | Double Dose
Number analyzed (Participants) | 5 | 6
participants
  Cough | 3 | 4
  Rhinorrhea | 3 | 3
  Shortness of breath | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Standard Dose | Double Dose
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 8/19 | 7/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Dose (N=19) | Double Dose (N=18)
Abdominal cramps (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Chest pain (General disorders) | 0 | 1
Feeling hot (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Tracheobronchitis (General disorders) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.